CLINICAL TRIAL: NCT02537353
Title: Prospective, Randomized Trial of Hemospray Plus Epinephrine Injection Versus Endoscopic Hemoclip Plus Epinephrine Injection in Nonvariceal Upper Gastrointestinal Bleeding
Brief Title: Trial of Hemospray Plus Epinephrine Injection Versus Endoscopic Hemoclip
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 14186713000000068
Record Dates: First submitted 2015-08-04; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-07

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Upper gastrointestinal bleeding; Hemospray; Endoscopic hemostasis
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — hemospray; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Placebo Comparator): Patients with a clinical diagnosis of upper gastrointestinal bleeding and that during endoscopy revealed to non-varicose bleeding lesions in the endoscopic treatment being necessary. The group will be submitted to injection of adrenaline at a proportion of 1: 10,000 in the four quadrants of the lesion associated with application of metal clips. The patients will be submitted to endoscopy exam in 12 to 24 hours after the therapeutic procedure to confirm the success of the therapy and measure if there the presence of rebleeding.
  Interventions: Device: Metal clips; Procedure: Endoscopy Exam; Drug: Adrenaline
- Group 2 (Active Comparator): Patients with a clinical diagnosis of upper gastrointestinal bleeding and that during endoscopy revealed to non-varicose bleeding lesions in the endoscopic treatment being necessary. The group will be submitted to injection of adrenaline at a proportion of 1: 10,000 in the four quadrants of the lesion associated with application adsorption powder, marketed under the name Hemospray. The patients will be submitted to endoscopy exam in 12 to 24 hours after the therapeutic procedure to confirm the success of the therapy and measure if there the presence of rebleeding.
  Interventions: Drug: Hemospray; Procedure: Endoscopy Exam; Drug: Adrenaline

INTERVENTIONS:
Device: Metal clips — The group will be shot of adrenaline 1: 10,000 in four quadrants, associated with application of metal clips.
  Arms: Group 1
Drug: Hemospray — The group will be shot of adrenaline 1: 10,000 in the four quadrants associated with application adsorption powder, marketed under the name Hemospray.
  Other Names: Dust adsorption
  Arms: Group 2
Procedure: Endoscopy Exam — All patients will be submitted to endoscopy exam in 12 to 24 hours after the therapeutic procedure to confirm the success of the therapy and measure if there the presence of rebleeding.
  Other Names: Upper Digestive Endoscopy
Drug: Adrenaline — The injection of adrenaline solution with 50% glucose at a proportion of 1: 10000 in four quadrants.

SUMMARY:
The non-variceal upper gastrointestinal bleeding is defined as gastrointestinal bleeding located proximal to the angle of Treitz, whose cause is not related to esophagogastric varices or gastropathy of portal hypertension.

Animal studies showed no absorption in the GIT and disposal within 48 hours of application, and no reported cases of obstruction. Recently, a prospective study involving 20 patients with upper gastrointestinal bleeding, showed that the application of hemospray ® promoted hemostasis in 95% of cases, confirmed by endoscopic revision 72h after application without any complication.

DETAILED DESCRIPTION:
The non-variceal upper gastrointestinal bleeding is defined as gastrointestinal bleeding located proximal to the angle of Treitz, whose cause is not related to esophagogastric varices or gastropathy of portal hypertension.

Despite all therapeutic guidelines and innovations introduced in recent decades, the incidence varies between 50 and 160 cases/100000 inhabitants / year and recent data show a mortality rate of approximately 10% in hospitalized patients. In the United States the upper gastrointestinal bleeding (HDA) promotes 300,000 hospitalizations per year.

The etiologies of non-variceal, HDA remains virtually unchanged over the past 20 years, peptic ulcer disease accounts for 40-50% of cases. Other less common causes are vascular ectasia, Mallory-Weiss lacerations, acute gastroduodenal mucosal lesions, Dieulafoy lesions, tumors and other rarer.

The HDA is manifested most often by hematemesis and / or melena. In a smaller proportion of patients can only be observed a drop in hemoglobin levels, and hemodynamic instability possible, without externalization of blood. There is also a smaller chance of rectal bleeding occur, which should indicate a bleeding of major consequence.

The management of patients with HDA should be systematized and as early as possible. Due to the unpredictability of the evolution of bleeding, all patients should be kept in the hospital environment and in the presence of hemodynamic and / or comorbidities should be considered high risk instability.

Hemodynamic stabilization is the initial step in the management of patients with HDA. Recent studies show that early and intensive resuscitation measures result in decreased length of hospitalization and mortality.

Following the hemodynamic maintenance, you should evaluate the presence of active bleeding, because when present, besides translating more severe, requiring a more rapid therapeutic intervention.

There are some findings predictive of severity of bleeding that can be evaluated from a clinical standpoint, they are: hemodynamic instability, need for continued transfusion, hematemesis with "fresh blood", rectal bleeding, bleeding that began during hospitalization, rebleeding during hospitalization in patients older than 60 years and presence of comorbidities.

Endoscopy (EDA) is the test of choice for the initial evaluation of bleeding of the upper digestive tract. The goals of endoscopic examination is to recognize the point of bleeding, hemostasis proceed when indicated and recognize stigma that suggest impending rebleeding. In peptic ulcers, using the classification of Forrest, the following findings are relevant: active arterial bleeding, visible vessel, and adherent clot. The risk of rebleeding these three groups without endoscopic treatment is estimated at 90%, 50% and 25%, respectively.

Endoscopic treatment has modified the natural evolution of non-variceal upper gastrointestinal bleeding. Several studies have shown that performing endoscopic therapy significantly reduces the risk of rebleeding and the length of hospital stay, need for surgical intervention and mortality.

Are risk factors for rebleeding: chronic renal failure, liver cirrhosis, low hemoglobin levels, the need for high doses of epinephrine for hemostasis and inexperienced endoscopist.

Endoscopic techniques in the treatment of existing HDA can be divided into three major groups: injection methods, thermal and mechanical.

In several clinical trials using two methods therapy (combination therapy) was more effective than using only one method.

The injection method is the use of sclerosing substances in the four quadrants of the lesion. The mechanism of action of hemostasis associated with the local tamponade, vasoconstriction and platelet aggregation. Among the available solutions for injection can be mentioned: adrenaline, ethanolamine, polidocanol, absolute ethanol and sodium chloride.

In the thermal heat production method causes protein denaturation tissue, collagen shrinkage and therefore obstruction of the vessel perivascular contraction. Thermal methods are used: Mono and bipolar electrocoagulation, argon plasma, laser and heater probe.

The treatment with mechanical methods has been developed in recent decades with the improvement of the devices used. In endoscopic practice who have proved effective are endoclipes and ligation.

The endoclip when compared to isolated therapeutic injection of adrenaline was superior in reducing rebleeding in peptic ulcers.

In a recent study, the use of argon plasma endoclip in ulcers with active bleeding were compared. The result demonstrated efficacy in both methods, no significant difference estastistica.

A new method developed for use in upper gastrointestinal bleeding and that proved to be safe and effective in clinical trials already done is dust adsorption (Hemospray ®). This new technology consists of a syringe containing the Hemospray ® powder, inorganic property comprises a group of minerals, highly adsorptive when in contact with blood, it becomes a cohesive powder and form a stable mechanical cap that covers the bleeding site. The powder is sprayed by means of a catheter connected to a container of carbon dioxide. The catheter tip should be positioned 1-2 cm from the site of bleeding and then short bursts of 1 to 2 seconds should be fired to stop the bleeding.

Studies in animals showed no absorption in the GIT and elimination within 48 hours of application, and no reported cases of obstruction. Recently, a prospective study involving 20 patients with upper gastrointestinal bleeding, showed that the application of hemospray ® promoted hemostasis in 95% of cases, confirmed by endoscopic revision 72h after application without any complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of upper gastrointestinal bleeding and that during endoscopy revealed to non-varicose bleeding lesions in the endoscopic treatment being necessary.

Exclusion Criteria:

* Pregnancy and History of endoscopic haemostatic procedure in the previous seven days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Initail hemostasis after endoscopic hemostatic procedure | up to 24 hours after endoscopic hemostatic procedure

SECONDARY OUTCOMES:
Rebleeding rate after endoscopic hemostatic procedure | participants will be followed for the duration of hospital stay, an expected avarage of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Felipe I Baracat, Study Chair — Hospital das Clínicas FMUSP; Eduardo GH de Moura, Principal Investigator — Hospital das Clínicas FMUSP